CLINICAL TRIAL: NCT03207971
Title: ANALISYS OF MULTIPLE GINGIVAL RECESSION TREATMENT WITH SUBEPITHELIAL CONNECTIVE TISSUE GRAFT REMOVED FROM PALATAL AREA WITH PREDOMINANCE OF LAMINA PROPRIA AND PREDOMINANCE OF SUBMUCOSA: CLINICAL EVALUATION AND LASER DOPPLER FLOWMETRY
Brief Title: ASSESSMENT OF CLINICAL PARAMETERS AND LASER DOPPLER FLOWMETRY FOR THE TREATMENT OF MULTIPLE GENGIVAL RECESSIONS WITH TWO TYPES OF SUBEPITELIAL CONNECTIVE GRAFT: RANDOMIZED CLINICAL STUDY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Rabelo Eustachio, Master of science student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10075100
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Gingival Recession, Generalized
Keywords: Gingival recession; Laser-Doppler Flowmetry; Periodontics
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCTG from palatal area with predominance of lamina propria (Active Comparator)
  Interventions: Procedure: Root coverage treatment with subepithelial connective tissue graft
- SCTG from palatal area with predominance of submucosa (Active Comparator)
  Interventions: Procedure: Root coverage treatment with subepithelial connective tissue graft

INTERVENTIONS:
Procedure: Root coverage treatment with subepithelial connective tissue graft — Periodontal plastic surgery aiming root coverage by palatal tissue graft removed from an area with predominance of lamina propria and predominance of submucosa.

SUMMARY:
Subepithelial connective tissue graft (SCTG) is considered the gold standard treatment for root coverage in Miller Class I and II single gingival recession. Therefore, scientific evidence is limited for multiple gingival recessions, only with extrapolation from single-tooth data. Depending on area and depth during the removal of the graft from palate, connective tissue presents different anatomic characteristics, geometric shapes and histological composition. Possibly different types of SCTGs present distinct volumetric stability and physiological process of revascularization. This randomized, split-mouth, double blind clinical trial aim to evaluate periodontal parameters (complete root coverage, gingival recession depth and width, gingival thickness, width of keratinized tissue, probing depth, clinical attachment, plaque and bleeding index) and gingival blood flow in recipient sites, comparing sites that received SCTG from palatal area with predominance of lamina propria and predominance of submucosa. Clinical measurements will be evaluated at baseline and 3, 6 and 12 months after surgical procedure. Blood flow flowmetry with laser doppler (LDF) will be analyzed at baseline and 3, 7,14 and 28 days after surgery. Participants will be invited to answer a questionnaire of aesthetic satisfaction and symptoms of pain and discomfort. Two experienced periodontists blind to experimental groups will be invited to observe the clinical outcomes and answer an aesthetic questionnaire. Data analysis will be performed by paired t-test if follow normal distribution or Wilcoxon if follow nonnormal distribution with significance level of 5% (p <0.05).

DETAILED DESCRIPTION:
This will be a randomized, double-blind, split-mouth clinical trial lasting 12 months. Participants will be selected from the Department of Periodontology of the Faculty of Dentistry of Bauru (FOB-USP). The sample will consist of systemically healthy individuals aged between 18 and 70 years. Patients will be included in the study if they meet the following inclusion criteria: (1) clinical diagnosis of multiple gingival recessions with at least one gingival recession ≥ 2 mm, including canines and premolars; (2) Miller class I and II gingival recession areas; (3) non-abrasive, erosive or carious root surfaces (4) unrotated, non-extruded and non-movable teeth (5) systemically healthy patients without contraindication to periodontal surgical procedures. The exclusion criteria will be: smokers, pregnant women, patients with a history of periodontal disease or recurrent abscess formation, patients previously submitted to surgical procedures for root coverage, patients taking anti-convulsant drugs, antihypertensives, contraceptives or immunosuppressors, patientes with low oral hygiene (plaque and bleeding index over 20%). The experimental protocol will be sent to the FOB-USP Human Research Ethics Committee for evaluation. Participants will receive detailed information about the study and will sign the Informed Consent Form after understanding all the steps of the research. All selected patients will be submitted to basic periodontal procedures (scaling, root planning, coronary polishing and oral hygiene instructions) before performing the surgical procedures. Patients should present plaque index and bleeding ≤ 20% throughout the study period.

Surgical Procedures

The experimental groups (A and B) will be treated through the association of subepithelial connective tissue graft (SCTG) and coronally advanced flap. Each individual will receive the types of treatment, randomly assigned to the right or left side. Group A will receive the submucosal predominant area for SCTG (removed from the anterior region of the lateral palate, more deeply) by the double-blade technique (Harris, 1997). This collection method allows a uniformity of the SCTG with standard thickness (1.5mm). Thus, the scalpel cable with double blades (1.5mm distance) will be used. The initial horizontal incision will be made on the palate, preserving 1-1.5 mm from the gingival margin of the teeth, until the complete deepening of the number 15C blades in the necessary extension previously defined for the receiving area. Internal vertical incisions will be performed for both sides of the horizontal incision and at the base of the graft to enable the SCTG removal. After the graft removal, the epithelial portion is extracted for subsequent stabilization of the graft to the recipient site.

Group B will be the one who will receive a graft whit a predominance of lamina propria (removed from the posterior region of the lateral palate, more superficially) by the technique of the deepithelialized graft. Two horizontal and two vertical incisions will be performed on the palate according to the extension needed for the recipient area, preserving 1-1.5 mm from the gingival margin of the teeth. These incisions will be made perpendicular to the palatine dome. Subsequently, for complete removal of the epithelial graft, an incision will be made with the 15 C blade, parallel to the palatal surface. The graft should be approximately 2 mm thick and after removal of the entire epithelium, the thickness should be 1.5 mm, measured with the anesthetic needle with endodontic stop and a digital pachymeter. The removal of the epithelium will be performed with the aid of reflector light (epithelium is firmer and more rugged and connective tissue, more flexible and soft) parallel to the surface of the graft. The difference in light reflection (epithelium reflects more than connective tissue) allows one to distinguish whether it has been removed (Zuchelli et al., 2010).

The width of the graft will be calculated according to the amount of tissue needed to cover the exposed roots plus mesial and distal 3mm and the amount of tissue required for the biopsy. The graft height will be the distance from the enamel cement junction (ECJ) to the buccal bone crest (Zuchelli et al., 2010). A small biopsy of the grafts (approximately 2mm x 6mm) will be removed for histomorphometric analysis. The donor area will be sutured with silk thread 4.0.

In the recipient areas, oblique incisions (from the ECJ to the gingival margin of the adjacent tooth) and intrasulcal incisions in the gingival recess defects will be performed with the objective of designing surgical papillae and anatomical papillae for the subsequent displacement of the flap to coronal (Zucchelli & DeSanctis, 2000). The incisions will be performed with a 15C scalpel blade and will extend to the adjacent teeth with gingival recessions. In the region of the interdental papilla, the deepithelialization will be performed with a scalpel blade. The flap will be of total thickness up to the height of the mucogingival junction to preserve greater thickness of flap that will be displaced on the bare root surface. In the most apical portion, the flap will be of partial thickness, eliminating muscular tensions and allowing greater mobility for subsequent accommodation of the flap by the same 2.5mm coronally to ECJ (Richardson et al, 2015). The root surfaces exposed to the buccal medium will be scraped with the aid of periodontal curettes.

After washing the recipient area with saline, SCTG with a standardized thickness of 1.5mm will be positioned over the exposed roots and sutured with 5-0 monofilament gluconate suture strands in adjacent connective tissue at the ECJ level. The flap will be advanced coronally so that each surgical papilla can be positioned over its respective anatomical papilla. In all cases, the ECJ and SCTG will be completely covered by the flap. With the same suture, sutures will be made to adapt the flap. The sutures will be removed 14 days after the surgical procedure. As a post-operative medication, all patients will receive analgesic, anti-inflammatory and instructed to gently wash the mouth with 0.12% chlorhexidine digluconate twice daily for 4 weeks. After the surgical procedure, patients will receive instructions on postoperative care verbally and also in writing. During this period they will be advised not to brush their teeth in the treated area. All patients will be followed weekly for 4 weeks, fortnightly for 6 months, and monthly for 12 months.

Clinical parameters:

Prior to the surgical procedure, all clinical measurements will be recorded by a calibrated examiner using computerized periodontal probe (Florida Probe®). Customized acrylic guides will be manufactured for each surgical area in order to allow successive measurements in the same position. The measurements will be rounded to the nearest 0.5 mm and repeated in the periods of 3, 6 and 12 months after surgery.

1. Depth of gingival recession (PR) - Distance in millimeters from ECJ to gingival margin at three points (mesial, center and distal);
2. Width of gingival recession (WGR) - Distance between interproximal gingival margins of the GR at the height of the most apical central portion of the JCE.
3. Clinical Probing Depth (CPD) - Distance in millimeters from the gingival margin to the bottom of the gingival sulcus at three points (mesial, center and distal);
4. Clinical attachment (CA) - Measured in mm from the bottom of the periodontal pocket to the cementoenamel junction at three sites per tooth (mesial, center and distal);
5. Width of keratinized mucosa (WKM) - Distance in millimeters from the gingival margin to the mucogingival junction at three points (mesial, center and distal).
6. Thickness of the keratinized mucosa (TKM): determined at 2mm apical the gingival margin at the central buccal site with anesthetic needle and endodontic stop and digital pachymeter (Paoloantonio et al., 2002, da Silva et al., 2004, Joly et al. 2007).
7. Plaque index (Ainamo and Bay, 1975): presence or absence of bacterial plaque on the 4 faces of the teeth (mesial, distal, buccal and lingual)
8. Bleeding index (Ainamo and Bay, 1975): presence or absence of bleeding after probing on the 4 faces of the teeth (mesial, distal, buccal and lingual)

Histomorphometric analysis of SCTG removed from the palate.

Although we can distinguish clinically the SCTG predominantly richer in lamina propria or submucosa, incisional biopsies of the grafts will be performed to confirm the nature of the tissue removed. The specimens will be approximately 2mm x 6mm being removed from the grafts of groups A and B. The specimens will be fixed in 10% formalin in phosphate buffer pH 7.3 for one week. They will then be rinsed in running water for 24 hours and kept in 70% ethanol until the next day. Histological processing will consist of dehydration in ethanol, diaphanization in xylol and inclusion in Histosec # (paraffin + synthetic resin) in an oven at 60oC. From the selected paraffin embedded cases, serial cuts with approximately 5 μm thickness will be performed, in a microtome; Then drawn in water and mounted on silanized slides. The cuts on the silanized slides will be submitted to routine histochemical technique staining with Hematoxylin and eosin.

Slides submitted to histochemical techniques will be evaluated with the aid of a microscope (CARL ZEISS, Germany). The first evaluation will determine if the epithelium has been completely removed. The second evaluation will be from the edge of the epithelial incision to the division that separates the lamina propria of the submucosa, measured in 5 different points. The total extent of the graft will be the sum of the last two measurements (Harris et al, 2003). All counts will be performed by a single calibrated examiner.

Laser-doppler flowmetry of the grafted area:

For the evaluation of the blood flow will be used the Laser Doppler Fluxometer (LDF) equipped with an infrared emitting diode laser (VMS-LDF2 DUAL CHANNEL- Laser Doppler Blood Flow and Temperature Monitor, trademark Moor instruments- FAPESP process number is 2012 / 13331-2). The maximum power of the diode laser is 2.5mW, emitting wavelengths in the order of 785nm ± 10nm. The time constant will be set to 0.1s and the bandwidth to 15kHz. It will be used 2 probes composed of 2 optical fibers of 0.25mm each, conditioned in an all steel of 1.5mm. The probes will be calibrated monthly in a solution that comes with the equipment kit.

Measurements with the LDF last 2 minutes. Three flow records of two points will be performed concomitantly with the interval of 1 minute between them. From these values, the average of the frequencies obtained will be considered to evaluate microvascularization at the determined points. There will be a total of 4 points evaluated by surgical field: two points at the base of the flap (alveolar mucosa immediately below the mucogingival junction) and two points at the border of the flap (two points at the margins of the gingiva).

Measurements with LDF in group A and B will be performed on the day of surgery before anesthesia and in the postoperative days of 3, 7, 14 and 28 days. To standardize the position (location and angulation) of the LDF probe relative to the gingival tissue at different evaluation times, the measurements will be performed with the aid of an individual acrylic guide supported on the tooth with perforations for fitting the point of the fiber optic probe (Donos et al., 2005; Retzepi M, 2007). In this way, the LDF probe will be inserted perpendicular to the tissues with a distance of 0.5 mm from the gingiva, remaining immobile during repeated measurements. In order to perform these measurements, patients will be comfortably accommodated in a standard semi-cline position, in the same dental chair, in a calm environment with a constant temperature (23 ± 20oC). Measurements will be performed by the same operator who has been properly calibrated and blinded to the experimental groups.

Subjective analyzes by questionnaires for patients and professionals:

Participants will be invited to answer a questionnaire with information about aesthetics, pain, discomfort, hygiene capacity of the area, sensitivity differences in donor areas. For this, analogue visual scales (AVS) will be used after 7, 14 and 28 days and at 3, 6 and 12 postoperative months. Likewise, the occurrence of adverse effects and /or postoperative complications will be documented.

Two experienced periodontists without the knowledge of the experimental groups will be asked to observe the clinical results after 7, 14 and 28 days and at the 3, 6 and 12 postoperative months and to answer a questionnaire including information about the healing pattern of the recipient and donor areas and aesthetics of the area.

Data Analysis

The sample estimate will be approximately 20 patients, and after a pilot study will be performed the sample calculation.

All examiners will be calibrated and the intraclass correlation coefficient will be calculated considering the parameters evaluated including clinical, microvascularization and histomorphometric analysis.

All individuals will receive the two treatments being randomly distributed to the right and left side. An independent statistician will generate a random sequence through software. During the surgical procedure, immediately after the preparation of the recipient surgical site, the investigator responsible for inclusion will open the opaque and sealed envelopes containing the information about the type of treatment that will receive on the right and left side.

The primary clinical outcome will be the depth of the gingival recession. The secondary clinical outcomes related to the tooth will be: (1) the complete root coverage (CRC) of the gingival recessions, (2) the width of the recession; (3) clinical attachment (CA); (4) clinical probing depth (CPD); (5) width and thickness of the keratinized mucosa (WKM, TKM); (6) analysis of microvascularization by LDF. The secondary clinical outcomes related to the patient will be: (1) aesthetic satisfaction; (2) pain and discomfort. Related to the specialist: (1) aesthetic satisfaction.

Descriptive statistics will be used to synthesize the data recorded in the initial and final evaluations. The statistical analysis of the clinical parameters will be performed to compare the initial values with the values after the experimental periods (6 and 12 months). The analysis of the data will be done by paired t test, if obeyed the distribution normal or Wilcoxon if it obeys the non-normal distribution. The level of significance adopted will be 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria: clinical diagnosis of multiple gingival recessions with at least one gingival recession ≥ 2 mm, including canines and premolars; (2) Miller class I and II gingival recession areas; (3) non-abrasive, erosive or carious root surfaces (4) unrotated, non-extruded and non-movable teeth (5) systemically healthy patients without contraindication to periodontal surgical procedures -

Exclusion Criteria:: smokers, pregnant women and infants, patients with a history of periodontal disease or recurrent abscess formation, patients previously submitted to surgical procedures for root coverage, patients taking anti-convulsant drugs, antihypertensives, contraceptives or immunosupressors, pacientes with low oral hygiene (plaque and bleeding index over 20%)

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-03 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Total root coverage measured with a periodontal probe in mm | One year
  Distance from cemento-enamel junction to gingival margin = 0 mm

SECONDARY OUTCOMES:
Keratinized mucosa width measured with a periodontal probe in mm | One year
  Ideal if keratinized mucosa width > 5mm

OTHER OUTCOMES:
Clinical Probing Depth | one year
  Distance in millimeters from the gingival margin to the bottom of the gingival sulcus at three points (mesial, center and distal). Ideal if <3mm
Clinical attachment | One year
  Measured in mm from the bottom of the periodontal pocket to the cemento-enamel junction at three sites per tooth (mesial, center and distal)
Thickness of the keratinized mucosa | One year
  Determined at 2mm apical the gingival margin at the central buccal site with anesthesic needle with endodontic stop and a digital pachymeter
Plaque index | One year
  Presence or absence of bacterial plaque on the 4 faces of the teeth (mesial, distal, buccal and lingual)
Bleeding index | One year
  Presence or absence of bleeding after probing on the 4 faces of the teeth (mesial, distal, buccal and lingual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuhr O, Baumer D, Hurzeler M. The addition of soft tissue replacement grafts in plastic periodontal and implant surgery: critical elements in design and execution. J Clin Periodontol. 2014 Apr;41 Suppl 15:S123-42. doi: 10.1111/jcpe.12185. PMID 24640997
- [Background] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963
- [Background] Chambrone L, Tatakis DN. Periodontal soft tissue root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S8-51. doi: 10.1902/jop.2015.130674. PMID 25644302